CLINICAL TRIAL: NCT04635956
Title: Anti-PD-1 Antibody Camrelizumab Combined With Cisplatin/Paclitaxel/Bevacizumab for Recurrent or Advanced Cervical Neuroendocrine Carcinomas: A Single Arm, Phase II Trial
Brief Title: Camrelizumab Combined With Chemotherapy for Recurrent or Advanced Cervical Neuroendocrine Carcinomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNET-PD1
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Chemotherapy; Anti-pd-1 Antibody; Cervical Neuroendocrine Carcinoma; Adverse Drug Event; Recurrent Cervical Carcinoma; Advanced Cervical Carcinoma; Objective Response Rate
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Uterine Cervical Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Intervention of platinum/etoposide/bevacizumab/camrelizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients will accept therapy consisting of platinum/etoposide/bevacizumab/camrelizumab
  Interventions: Drug: Drug therapy

INTERVENTIONS:
Drug: Drug therapy — 6 courses of platinum/etoposide/bevacizumab/camrelizumab and a total period of 12 months bevacizumab/camrelizumab

SUMMARY:
Recurrent or advanced cervical neuroendocrine carcinoma (NEC) is refractory to multimodal treatment, even to extensive therapy. Chemotherapy, consisting of platinum and etoposide, remains the main therapy for recurrent or advanced cervical NEC. In addition, bevacizumab has shown progression-free benefits in recurrent or advanced cervical cancer. Case report suggested anti-PD-1 antibody may have antitumor activities in NEC. Based on these evidences, a phase 2, single arm trial is conducted to explore the objective response rate (ORR) of platinum/etoposide/bevacizumab/anti-PD-1 antibody (camrelizumab) for the treatment of recurrent or advanced cervical NEC. This trial is to enroll 20 patients, who would accept 6 courses of platinum/etoposide/bevacizumab/camrelizumab. If the patient achieved complete or partial remission, a total period of 12 months bevacizumab/camrelizumab will be given as maintain therapy. The primary endpoint is ORR. The second endpoints are severe adverse events according to criteria of Common Terminology Criteria for Adverse Events (CTCAE) and iRECIST Guideline, and critical changes of laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed recurrent or advanced cervical neuroendocrine carcinoma
* Aged 18 years or older
* No immunosuppressive disease
* Signed an approved informed consents
* Performance status of ECOG 0-1

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 1 years
  proportion of partial or complete remission after intervention

SECONDARY OUTCOMES:
severe adverse events | 1 year
  grade 3/4 adverse events and mortality according to criteria of Common Terminology Criteria for Adverse Events (CTCAE) and iRECIST Guideline
a composite changes of important laboratory testing | 1 year
  these changes include liver/kidney/myocardiac functions, insulin resistance, functions of adrenal gland

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China